CLINICAL TRIAL: NCT03046420
Title: Hypertension Prevalence, Treatment Patterns and Outcomes in Long-Term Care Facilities
Brief Title: Hypertension in Long-Term Care Facilities
Status: Completed | Type: Observational
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Erwin A. Aguilar, Associate Professor, Louisiana State University Health Sciences Center in New Orleans
Other Study IDs: LSUIRB 9571
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Chart review — This is a retrospective chart review study. The charts of patients who meet the inclusion criteria will be abstracted into a standardized electronic case report form, as described in Section 5. A standardized case report form for each patient will be created so as to collect uniform data. Charts data for one year back to the start date of data abstraction will be included in the study

SUMMARY:
This study is exploratory in nature and seeks to describe hypertension diagnosis and management among patients in long-term care (LTC) facilities.

Specifically, the primary objective is to:

• Identify LTC patients who are diagnosed with hypertension and assess the management and different outcomes of proper control of BP regarding to incidence of falls, cognitive decline, kidney diseases, cardiovascular diseases and incidence of cerebrovascular accidents

The secondary objectives are to:

Describe treatment patterns of hypertension in LTC facilities

* Identify patients who are receiving non-pharmacological treatment and effectiveness of this modality of treatment.
* Identify different classes of drugs used to treat hypertension in patients staying at LTC facility
* Identify different drug adverse effects encountered by patients receiving medical treatment.
* Identify patients who achieved normal blood pressure according to current guidelines

DETAILED DESCRIPTION:
Isolated systolic hypertension is more common in elderly than younger adults. Also blood pressure (BP) in elderly tends to be very high, difficult to treat. Many studies are done to understand the mechanism of hypertension in older adults, most of them concluded that the main mechanisms are chronic inflammation, oxidative stress and endothelial dysfunction. Hypertension is often called a "silent killer" and it is a major high risk factor of heart, chronic kidney and cerebrovascular diseases . Systolic BP (SBP) gradually increases from early adulthood to old age, whilst diastolic BP (DBP) increases until around 50 years of age then reaches a plateau before decreasing again , causing widening of pulse pressure, and elevated blood pressure known as Isolated Systolic Hypertension (ISH).

There is a general consensus across international guidelines for a recommended target BP of SBP ≤ 140 mmHg and DBP≤90 mmHg for the general adult population without diabetes mellitus (DM) however the treatment of hypertension in the elderly requires further clarification and further studies as many international guidelines are inconsistent in providing recommendation on optimal BP for both initiation ant of therapy ad for treatment in the elderly due to the limited outcome date form randomized controlled trials (RCT) in this population .

The American Heart Association recommendations to initiate treatment starting with lifestyle changes and then medication if necessary at 140/90 mmHg until age 80, then at 150/90 mmHg for adults ˃ 80 years old '

The 2014 Joint National Committee's eights report (JNC 8) recommends that in general population aged ≥60 years, to initiate pharmacologic treatment to lower BP at systolic BP (SBP) ≥150 mm Hg or diastolic BP (DBP) ≥90 mm Hg and treat to a goal SBP<150 mm Hg and goal DBP <90 mm Hg . However Reisin et al published a commentary on JNC 8 disagreeing with it, having a concern that increasing the SBP level requiring treatment in those ≥60 years old to ≥150/≥90 mmHg may adversely affect renal function.

As Per the European society of Cardiology and the European Society of Hypertension: in elderly patients drug treatment is recommended when systolic BP is ≥160 mmHg, or ≥140 mmHg if younger than 80 years and treatment is well tolerated. It is not recommended to initiate antihypertensive treatment at high normal BP and in younger patients with isolated systolic hypertension.

As per 2011 NICE guidelines the aim for target average blood pressure is <135/85 mmHg for People <80 years old and <145/85mmHg for people ≥80 years .

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with hypertension
* Be ≥ 60 years of age
* Stays at the LTC facility for at least 3 months

Exclusion Criteria:

* Patients under age of 60 Patients without diagnosis of hypertension Terminally ill patients and hospice patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study population will consist of patients residing at a LTC facility affiliated with Louisiana State University Health Sciences Center in New Orleans (LSUHSC-NO) at the start of data collection for a minimum of three months period. Chart and claims data will be collected retrospectively back to one year from date of the start date of data abstraction.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Management of Hypertension | 1 year
  outcomes of proper control of blood pressure regarding to incidence of falls, cognitive decline, kidney diseases, cardiovascular diseases and incidence of cerebrovascular accidents

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Aguilar, PharmD, MPH, Principal Investigator — LSU Health Sciences Center in New Orleans
Locations (1):
- LSU Health Sciences Center, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ostchega Y, Dillon CF, Hughes JP, Carroll M, Yoon S. Trends in hypertension prevalence, awareness, treatment, and control in older U.S. adults: data from the National Health and Nutrition Examination Survey 1988 to 2004. J Am Geriatr Soc. 2007 Jul;55(7):1056-65. doi: 10.1111/j.1532-5415.2007.01215.x. PMID 17608879
- [Background] Butt DA, Harvey PJ. Benefits and risks of antihypertensive medications in the elderly. J Intern Med. 2015 Dec;278(6):599-626. doi: 10.1111/joim.12446. Epub 2015 Oct 26. PMID 26497967
- [Background] Franklin SS, Jacobs MJ, Wong ND, L'Italien GJ, Lapuerta P. Predominance of isolated systolic hypertension among middle-aged and elderly US hypertensives: analysis based on National Health and Nutrition Examination Survey (NHANES) III. Hypertension. 2001 Mar;37(3):869-74. doi: 10.1161/01.hyp.37.3.869. PMID 11244010
- [Background] Buford TW. Hypertension and aging. Ageing Res Rev. 2016 Mar;26:96-111. doi: 10.1016/j.arr.2016.01.007. Epub 2016 Feb 1. PMID 26835847
- [Background] Franklin SS. Hypertension in older people: part 1. J Clin Hypertens (Greenwich). 2006 Jun;8(6):444-9. doi: 10.1111/j.1524-6175.2006.05113.x. PMID 16760685
- [Background] Franklin SS, Gustin W 4th, Wong ND, Larson MG, Weber MA, Kannel WB, Levy D. Hemodynamic patterns of age-related changes in blood pressure. The Framingham Heart Study. Circulation. 1997 Jul 1;96(1):308-15. doi: 10.1161/01.cir.96.1.308. PMID 9236450
- [Background] Kjeldsen S, Feldman RD, Lisheng L, Mourad JJ, Chiang CE, Zhang W, Wu Z, Li W, Williams B. Updated national and international hypertension guidelines: a review of current recommendations. Drugs. 2014 Nov;74(17):2033-51. doi: 10.1007/s40265-014-0306-5. PMID 25315030
- [Background] Go AS, Bauman MA, Coleman King SM, Fonarow GC, Lawrence W, Williams KA, Sanchez E. An effective approach to high blood pressure control: a science advisory from the American Heart Association, the American College of Cardiology, and the Centers for Disease Control and Prevention. J Am Coll Cardiol. 2014 Apr 1;63(12):1230-1238. doi: 10.1016/j.jacc.2013.11.007. Epub 2013 Nov 15. No abstract available. PMID 24246165
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Reisin E, Harris RC, Rahman M. Commentary on the 2014 BP guidelines from the panel appointed to the Eighth Joint National Committee (JNC 8). J Am Soc Nephrol. 2014 Nov;25(11):2419-24. doi: 10.1681/ASN.2014040371. Epub 2014 Aug 11. PMID 25114277
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F, Redon J, Dominiczak A, Narkiewicz K, Nilsson PM, Burnier M, Viigimaa M, Ambrosioni E, Caufield M, Coca A, Olsen MH, Schmieder RE, Tsioufis C, van de Borne P, Zamorano JL, Achenbach S, Baumgartner H, Bax JJ, Bueno H, Dean V, Deaton C, Erol C, Fagard R, Ferrari R, Hasdai D, Hoes AW, Kirchhof P, Knuuti J, Kolh P, Lancellotti P, Linhart A, Nihoyannopoulos P, Piepoli MF, Ponikowski P, Sirnes PA, Tamargo JL, Tendera M, Torbicki A, Wijns W, Windecker S, Clement DL, Coca A, Gillebert TC, Tendera M, Rosei EA, Ambrosioni E, Anker SD, Bauersachs J, Hitij JB, Caulfield M, De Buyzere M, De Geest S, Derumeaux GA, Erdine S, Farsang C, Funck-Brentano C, Gerc V, Germano G, Gielen S, Haller H, Hoes AW, Jordan J, Kahan T, Komajda M, Lovic D, Mahrholdt H, Olsen MH, Ostergren J, Parati G, Perk J, Polonia J, Popescu BA, Reiner Z, Ryden L, Sirenko Y, Stanton A, Struijker-Boudier H, Tsioufis C, van de Borne P, Vlachopoulos C, Volpe M, Wood DA. 2013 ESH/ESC guidelines for the management of arterial hypertension: the Task Force for the Management of Arterial Hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). Eur Heart J. 2013 Jul;34(28):2159-219. doi: 10.1093/eurheartj/eht151. Epub 2013 Jun 14. No abstract available. PMID 23771844
- [Background] Jaques H; National Institute for Health and Clinical Excellence (NICE). NICE guideline on hypertension. Eur Heart J. 2013 Feb;34(6):406-8. No abstract available. PMID 23520636
- [Background] Weber MA, Schiffrin EL, White WB, Mann S, Lindholm LH, Kenerson JG, Flack JM, Carter BL, Materson BJ, Ram CV, Cohen DL, Cadet JC, Jean-Charles RR, Taler S, Kountz D, Townsend R, Chalmers J, Ramirez AJ, Bakris GL, Wang J, Schutte AE, Bisognano JD, Touyz RM, Sica D, Harrap SB. Clinical practice guidelines for the management of hypertension in the community a statement by the American Society of Hypertension and the International Society of Hypertension. J Hypertens. 2014 Jan;32(1):3-15. doi: 10.1097/HJH.0000000000000065. No abstract available. PMID 24270181
- [Background] Stevens PE, Levin A; Kidney Disease: Improving Global Outcomes Chronic Kidney Disease Guideline Development Work Group Members. Evaluation and management of chronic kidney disease: synopsis of the kidney disease: improving global outcomes 2012 clinical practice guideline. Ann Intern Med. 2013 Jun 4;158(11):825-30. doi: 10.7326/0003-4819-158-11-201306040-00007. PMID 23732715
- [Background] Dasgupta K, Quinn RR, Zarnke KB, Rabi DM, Ravani P, Daskalopoulou SS, Rabkin SW, Trudeau L, Feldman RD, Cloutier L, Prebtani A, Herman RJ, Bacon SL, Gilbert RE, Ruzicka M, McKay DW, Campbell TS, Grover S, Honos G, Schiffrin EL, Bolli P, Wilson TW, Lindsay P, Hill MD, Coutts SB, Gubitz G, Gelfer M, Vallee M, Prasad GV, Lebel M, McLean D, Arnold JM, Moe GW, Howlett JG, Boulanger JM, Larochelle P, Leiter LA, Jones C, Ogilvie RI, Woo V, Kaczorowski J, Burns KD, Petrella RJ, Hiremath S, Milot A, Stone JA, Drouin D, Lavoie KL, Lamarre-Cliche M, Tremblay G, Hamet P, Fodor G, Carruthers SG, Pylypchuk GB, Burgess E, Lewanczuk R, Dresser GK, Penner SB, Hegele RA, McFarlane PA, Khara M, Pipe A, Oh P, Selby P, Sharma M, Reid DJ, Tobe SW, Padwal RS, Poirier L; Canadian Hypertension Education Program. The 2014 Canadian Hypertension Education Program recommendations for blood pressure measurement, diagnosis, assessment of risk, prevention, and treatment of hypertension. Can J Cardiol. 2014 May;30(5):485-501. doi: 10.1016/j.cjca.2014.02.002. Epub 2014 Feb 22. PMID 24786438
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] Prevention of stroke by antihypertensive drug treatment in older persons with isolated systolic hypertension. Final results of the Systolic Hypertension in the Elderly Program (SHEP). SHEP Cooperative Research Group. JAMA. 1991 Jun 26;265(24):3255-64. PMID 2046107
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272